CLINICAL TRIAL: NCT03970889
Title: Pilot Study to Test Efficacy of Real-time Reminders on Apple Watch To Decrease Late or Missed Meal Boluses
Brief Title: Real-time Reminders To Decrease Late or Missed Meal Boluses
Acronym: Klue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Bruce Buckingham, Professor of Pediatric Endocrinology, Stanford University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 47137
Record Dates: First submitted 2018-08-23; First posted 2019-06-03 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Type1 Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Subjects are randomized so that half will use the Klue App in the first 6 weeks of the study, and half will use the Klue App during the second 6 weeks of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (No Intervention): Participants will be in their usual care, wearing a continuous glucose sensor and taking insulin by pump or by pens with memory
- Klue (Experimental): Subjects will wear an Apple watch on their dominant hand and receive alerts when eating behavior is detected by the Klue software.
  Interventions: Device: Klue

INTERVENTIONS:
Device: Klue — Klue is a software program the uses an Apple watch to detect hand motions which are indicative of eating.
  Arms: Klue

SUMMARY:
This study is examining whether the Klue app is effective in detecting missed or late meal boluses in patients with Type 1 diabetes. The app is programmed onto an Apple Watch and will detect potential missed boluses from hand motion. It will send text alerts to the user asking if they have bolused. This is a pilot study and will assess whether there is a change in the number of missed meal boluses in the two weeks prior to each visit. If the findings are significant, this software can be integrated in future closed-loop algorithms for automatic insulin delivery.

DETAILED DESCRIPTION:
This will be a randomized, cross-over, unblinded study with subjects randomized upon entry into the study to either begin using the Klue software for 6 weeks or to continue with their usual care for 6 weeks. Subjects are eligible for enrollment if they are using a continuous glucose monitor (CGM) and insulin pumps or an insulin pen with memory and CGM, are missing or late in giving at least 4 food boluses in the previous two weeks, and they have an iPhone. Missing or late meal boluses will be assessed through their pump/pen and sensor downloads. This is a pilot study. The investigators do not have preliminary data to do a true power calculation. The primary outcome will be the change in the number of missed meal boluses in the two weeks prior to each visit. Secondary outcome measures will be the number of missed meal boluses in each month of the study, change in HbA1c levels (measured every 6 weeks), accuracy of the Klue software in detecting meals (true positive and false positive rates), and a user satisfaction survey.

ELIGIBILITY:
Inclusion Criteria:

1. Age 13 and over
2. On an insulin pump for at least 3 months and using CGM or using an insulin pen with memory and a CGM
3. Willing to wear a CGM at least 70% of the time while in the study
4. Using an iPhone
5. Willing to wear an Apple watch on their dominant hand while awake
6. Missing or late in giving at least four food boluses in the previous two weeks
7. Understanding and willingness to follow the protocol and sign informed consent
8. Ability to speak, read and write in the language of the investigators

Exclusion Criteria:

1. Pregnant or lactating
2. A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol
3. Current treatment for a seizure disorder
4. Inpatient psychiatric treatment in the past 6 months

Note: Adequately treated thyroid disease and celiac disease do not exclude subjects from enrollment. They may be participating in another trial, if this study is approved by the investigators of the other trial.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-10-12 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Change in the number of missed meal boluses | The two weeks prior to each study visit
  A missed meal bolus is defined by no insulin dose within 2 hours from the start of the CGM rise.

SECONDARY OUTCOMES:
Change in time in range | data for 1 month prior to each study visit at baseline, 6 weeks and 12 weeks of this 12 week study for each subject
  sensor glucose values between 70-180 mg/dl
Positive predictive value of a Klue meal alert | All data for the 6 weeks on the Klue intervention arm when Klue is active
  Percent of time a meal alert signaled a meal

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Buckingham, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burdick J, Chase HP, Slover RH, Knievel K, Scrimgeour L, Maniatis AK, Klingensmith GJ. Missed insulin meal boluses and elevated hemoglobin A1c levels in children receiving insulin pump therapy. Pediatrics. 2004 Mar;113(3 Pt 1):e221-4. doi: 10.1542/peds.113.3.e221. PMID 14993580
- [Background] Olinder AL, Kernell A, Smide B. Missed bolus doses: devastating for metabolic control in CSII-treated adolescents with type 1 diabetes. Pediatr Diabetes. 2009 Apr;10(2):142-8. doi: 10.1111/j.1399-5448.2008.00462.x. Epub 2008 Oct 24. PMID 19175898